CLINICAL TRIAL: NCT05023408
Title: Intralesional Bleomycin Versus Cryotherapy for Treatment of Cutaneous Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Javaria Rahmatullah, FCPS II Postgraduate Trainee, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JinnahPMC
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Cutaneous Warts
Keywords: cutaneous warts,intralesional bleomycin,cryotherapy,efficacy
MeSH Terms: interventions — Bleomycin; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralesional Bleomycin (Experimental): Intralesional Bleomycin has been given to palmo plantar warts. Generic name: Bleomycin Dose: 1mg/1ml (0.1%) Frequency: every 2 weekly for 6 weeks.
  Interventions: Drug: Bleomycin Injection
- Cryotherapy (Experimental): Cryotherapy has been given to palmo plantar warts. Frequency: every 2 weekly for 6 weeks
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Drug: Bleomycin Injection — Intralesional Bleomycin used for treatment of cutaneous warts.
  Other Names: Bleomycin Sulfate
  Arms: Intralesional Bleomycin
Procedure: Cryotherapy — Cryotherapy used for comparison of efficacy.
  Arms: Cryotherapy

SUMMARY:
The purpose of the study was to determine the efficacy of intralesional bleomycin in comparison to cryotherapy on participants having cutaneous warts.

DETAILED DESCRIPTION:
This study was conducted in the Department of Dermatology of Jinnah Postgraduate Medical Centre, Karachi from January to June 2021 after receiving approval from the institutional ethical and research committee of hospital.

Sample size was calculated through NCSS software. Total of one fifty four non-admitted patients were assigned two study groups with equal sample size of 77 randomly through lottery method. Those patients aged between 18 to 60 years of either gender with cutaneous warts for > 1 week to 48 weeks were included after written informed consent. Patients treated previously for warts by any methodology, with history of vascular disease, immunocompromised, hypertension, cardiovascular disorder, pregnancy, lactation and hypersensitivity to lidocaine were excluded.

All demography, clinical history was recorded by a principal investigator on a predesigned Performa , informed written consent was taken before enrolment.

Group A received intralesional bleomycin 0.1% therapy until the lesion blanched. It was prepared manually by diluting 15 mg powder in 5 ml distilled water and then each ml was further diluted by adding 2ml of 2% lignocaine, double the amount taken from the vial, so that concentration became 1mg/1ml (0.1%). Group B patients were treated with liquid nitrogen with the help of a cotton swab wrapped on a wooden stick and was applied firmly with 01 mm extra healthy skin margin until the lesion blanched.

Follow-up was carried out at 02, 04 and 06 weeks. Both the groups were assessed and compared for efficacy after 6 weeks of therapy. SPSS 23 was used for analyzing data.

ELIGIBILITY:
Inclusion Criteria:

* • Age18 to 60 years

  * Either gender.
  * Diagnosed cases of cutaneous warts as per operational definition for > 1 week to 48 weeks.

Exclusion Criteria:

* • Previously treated for warts by any methodology, assessed by history and clinically.

  * Patients with hypertension, cardiovascular disorder, pregnancy, lactation, vascular diseases, assessed by history, clinically & by positive autoimmune profile.
  * Hypersensitivity to lidocaine.
  * No given informed written consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
change in morphology of cutaneous warts. | 6 weeks
  There is complete remission of cutaneous warts, assessed clinically

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ghafoor, FCPS, Study Director — Jinnah Postgraduate Medical Centre
Locations (1):
- Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No